CLINICAL TRIAL: NCT06329414
Title: Acceptability and Feasibility of Transcranial Magnetic Stimulation (TMS) for Depression in Multiple Sclerosis
Status: Recruiting | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Kathleen Shangraw, Resident Physician, University of Utah
Other Study IDs: 00164631
Record Dates: First submitted 2024-03-15; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Multiple Sclerosis; Major Depressive Disorder; Treatment Resistant Depression
Keywords: multiple sclerosis; depression; major depressive disorder; treatment resistant depression; transcranial magnetic stimulation; TMS
MeSH Terms: conditions — Multiple Sclerosis; Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant; Depression

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The goal of this single-arm, observational pilot study is to learn about the safety, feasibility, preliminary efficacy of TMS for the treatment of depression in people with MS. Participants will receive outpatient TMS treatment over the course of 5-6 weeks. Participants will complete validated questionnaires and exams before, during, and after treatment.

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic, immune-mediated disease of the central nervous system. Depression, or major depressive disorder, is highly prevalent in people with MS and often has a serious impact on quality of life. MDD can be difficult to treat with medications in MS. Transcranial magnetic stimulation (TMS) is a safe and approved treatment for treatment-resistant depression in the general population. However, little is known about the use of TMS for MDD in people with MS. This pilot study will evaluate the safety, feasibility, and preliminary efficacy of TMS for MDD in MS. Participants will receive outpatient neuronavigated-TMS for MDD. Various measures of MS and MDD symptoms will be monitored over the course of treatment. Clinical brain imaging will also be compared before and after TMS.

ELIGIBILITY:
Inclusion Criteria:

* Established diagnosis of multiple sclerosis (any subtype) by 2017 McDonald criteria
* Established diagnosis of major depressive disorder (MDD) by DSM-5 criteria
* Eligible for transcranial magnetic stimulation (rTMS) for depression

Exclusion Criteria:

* MS relapse and/or steroid use within 3 months
* Active suicidal ideation
* History of seizure/epilepsy, brain tumor, or stroke
* History of bipolar disorder or psychosis
* Currently or planning to become pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults diagnosed with MDD and MS who are eligible for TMS
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2024-01-16 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of TMS treatment for MDD, per participant retention rates. | 10 weeks
Safety and tolerability, to be evaluated by side effects and adverse events over the course of treatment. | 10 weeks

SECONDARY OUTCOMES:
Depression response rates (50% reduction in symptoms) will be measured using MADRS scores before and after treatment. | 10 weeks
Depression remission rates will be measured using MADRS scores before and after treatment. | 10 weeks
MS lesion burden on MRI will be compared before and after treatment to determine impact of TMS on white matter disease burden. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah Health, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No